CLINICAL TRIAL: NCT00554476
Title: Comparison of Two Combined Therapeutic Methods for Treatment of Lateral Epicondylitis: A Randomized Clinical Trial
Brief Title: Comparison of Two Combined Therapeutic Methods for Treatment of Lateral Epicondylitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Because the sample volume was completed during three years.
Sponsor: Azad University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT-246910-06
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2007-11-07 (Estimated); Status verified 2007-11

CONDITIONS: Lateral Epicondylitis
Keywords: Lateral Epicondylitis; Treatment; Corticosteroid; Elbow Cast; Icing; NSAIDs
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Triamcinolone Acetonide- Indomethacin-Cryotherapy-Casting

SUMMARY:
To compare the effectiveness of two combined therapeutic methods including corticosteroid injections with elbow cast versus ice massage and non-steroidal anti inflammatory drugs (NSAIDs).

DETAILED DESCRIPTION:
Design: Randomized clinical trial. Setting: Boo-Ali and Baqyiatallah Hospital in Tehran. Patients: 50 randomly selected patients, in two groups of 25 subjects. Interventions: Corticosteroid injections with elbow cast versus icing and NSAIDs.

Outcome measures: Patients were evaluated for outcomes, complications and patients' satisfaction at 2nd, 4th, and 12th week after beginning of treatment. We measured the pain severity by Visual Analogue Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* pain at the lateral side of the elbow
* pain at the lateral epicondyle during resisted dorsiflexion of the wrist with the elbow in full extension, or resisted extension of middle finger at the metacarpophalangeal joint
* pain to be continued for longer than 6 weeks or even with recurrent pain during similar period

Exclusion Criteria:

* previous history of receiving any treatment for lateral epicondylitis within 6 months prior to intervention
* patients who were unable to return for follow up
* patients with nerve entrapment
* pregnancy
* breast-feeding
* presence of systemic neuromuscular disorders such as myasthenia gravis
* upper limb fractures
* other arm/forearm pathology such as radial nerve compression
* known thrombocytopenia
* coagulopathy or bleeding diathesis
* history of diffuse pain syndrome
* history of inflammatory arthropathy
* intolerance/allergy to corticosteroids or NSAIDs or any contraindication for these
* untreated depression
* history of narcotic use for pain management greater than 1 month or history of narcotic abuse problem

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-01; Study Completion 2006-04

PRIMARY OUTCOMES:
visual analogue scale (VAS)

SECONDARY OUTCOMES:
Patient's satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Jaleh Hassanloo, MD, Principal Investigator — Department of Orthopedics, Boo-Ali Hospital
Locations (1):
- Azad University of Medical Sciences, Boo-Ali Hospital, Tehran, Tehran Province, Iran